CLINICAL TRIAL: NCT04606030
Title: LymphBridge: Prospective Evaluation of the BioBridge Scaffold as an Adjunct to Lymph Node Transplant for Upper Extremity Lymphedema
Brief Title: LymphBridge: Surgical Evaluation for Breast Cancer-Associated Lymphedema (BioBridge)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fibralign Corporation (Industry)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R44CA203608 (NIH)
Record Dates: First submitted 2020-10-25; First posted 2020-10-28 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Lymphedema; Edema
Keywords: Lymphedema; Edema
MeSH Terms: conditions — Lymphedema; Edema

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, control arm
Who Masked: Outcomes Assessor
Masking Description: Partially Blinded: Patients will be informed which group they are randomized into and given the option to opt out of the study. Investigators (other than surgeons conducting surgery) and study personnel involved in patient measurements will be unaware of the patient treatment option.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- BioBridge treatment group (Experimental): Vascularized Lymph Node Transplant surgery (VLNT) supplemented by BioBridge Collagen Matrix implantation
  Interventions: Device: BioBridge® Collagen Matrix; Procedure: Vascularized Lymph Node Transfer (VLNT)
- Control group (Active Comparator): Vascularized Lymph Node Transplant surgery (VLNT) only
  Interventions: Procedure: Vascularized Lymph Node Transfer (VLNT)

INTERVENTIONS:
Device: BioBridge® Collagen Matrix — BioBridge Collagen Matrix (BioBridge) is a sterile implantable bio-compatible and biodegradable surgical mesh ribbon comprised of highly purified porcine collagen. The Class II device was cleared by CDRH Division of Surgical Devices on 8 January 2016 under 510(k) K151083. The device will be used for soft tissue surgical support at the time of vascularized lymph node transplant surgery (VLNT); the device will be used, specifically, for surgical support of the lymphatic component of the soft tissue.
  Arms: BioBridge treatment group
Procedure: Vascularized Lymph Node Transfer (VLNT) — Micro-surgical procedure for vascularized lymph node transfer (VLNT)

SUMMARY:
To investigate whether the addition of Fibralign's BioBridge® Collagen Matrix (BioBridge) devices to the standard surgery for vascularized lymph node transfer will improve the outcome of surgical treatment in lymphedema of the upper arm.

DETAILED DESCRIPTION:
The proposed study utilizes Fibralign's BioBridge® Collagen Matrix (BioBridge), a sterile implantable biocompatible and biodegradable surgical mesh ribbon comprised of highly purified porcine collagen. The Class II device was cleared by CDRH Division of Surgical Devices on 8 January 2016 under 510(k) K151083. The device will be used for soft tissue surgical support at the time of vascularized lymph node transplant surgery (VLNT); the device will be used, specifically, for surgical support of the lymphatic component of the soft tissue.

Primary endpoint is the post surgical % change in excess limb volume, measured at 12 months following the surgical procedure.

Secondary endpoints are change in quality of life scores measured by LLIS and change in lymphatic function as measured by indocyanine green (ICG) fluorescence imaging.

ELIGIBILITY:
Inclusion Criteria:

The subject must be a breast cancer survivor, at least 3 years beyond completion of cancer therapy, free of clinical disease, and eligible for surgical intervention. Participants who are not able to safely undergo general anesthesia and/or perioperative care for VLNT are excluded.

* Ages 18 to 75 years (inclusive)
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
* Life expectancy > 2 years
* Acquired (secondary) upper limb lymphedema secondary to breast cancer treatment
* The participant must be eligible for surgical intervention
* Swelling of 1 limb that is not completely reversed by elevation or compression
* Stage I-II lymphedema at screening, based on the International Society of Lymphology (ISL) staging system
* Participants must have no evidence of disease (NED), have completed breast cancer therapy 3 years prior to enrollment; use of endocrine therapy is allowed.
* Completion of a full course of complete decongestive therapy (CDT), according to ISL guidelines at least 12 weeks prior to screening, including use of compression garments for at least 12 weeks without change in regimen
* Willingness to comply with recommended regimen of self care, with consistent use of compression garments from screening through the entire study duration (through the safety follow up visit), excluding the first 3 weeks postoperatively where patients are required to not wear compression. Self bandaging, use of nighttime compression garments, and intermittent pneumatic compression devices are allowed, but the procedures and regimens are expected to remain consistent from screening though the entire study duration.
* Consistent use of an appropriately sized compression garment for daytime use.
* Limb volume (LV) in the affected limb and unaffected limb must be at least 10% of each other.
* Evidence of abnormal bioimpedance ratio, if feasible, based upon unilateral disease: L Dex > 10 units.
* Willingness and ability to comply with all study procedures, including measurement of skin biopsy, and preoperative and postoperative imaging studies.
* Willingness and ability to understand, and to sign a written informed consent form document

Exclusion Criteria:

* Edema arising from increased capillary filtration will be excluded (venous incompetence).
* Inability to safely undergo general anesthesia and/or perioperative care related to vascularized lymph node transfer
* Concurrent participation in a clinical trial of any other investigational drug or therapy, regardless of indication, within 1 month before screening or 5 times the drug's half life, whichever is longer
* Recent initiation (≤ 12 weeks) of CDPT for lymphedema
* Other medical condition that could lead to acute limb edema, such as (but not limited to) acute venous thrombosis or heart failure
* Other medical condition that could result in symptoms overlapping those of lymphedema in the affected limb (eg, pain, swelling, decreased range of motion)
* History of clotting disorder (hypercoagulable state)
* Chronic (persistent) infection in the affected limb
* Infection of the lymphedema limb within 1 month prior to screening
* Currently receiving chemotherapy or radiation therapy
* Current evidence, or a history of malignancy within the past 3 years (except for non melanoma skin cancer or cervical cancer in situ treated with curative intent). If the participant has undergone cancer treatment, this must have been completed > 3 years prior to enrollment.
* Significant or chronic renal insufficiency (defined as serum creatinine > 2.5 mg/dL or an estimated glomerular filtration rate [eGFR] < 30 mL/min at screening) or requires dialytic support
* Hepatic dysfunction, defined as alanine transaminase (ALT) or aspartate transaminase (AST) levels > 3 × upper limit of the normal range (ULN) and/or bilirubin level > 2 × ULN at screening
* Absolute neutrophil count < 1500 mm3 at screening
* Hemoglobin concentration < 9 g/dL at screening
* Body Mass Index (BMI) >35
* Known sensitivity to porcine products
* Anaphylaxis to iodine
* Pregnancy or nursing
* Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening
* Any reason (in addition to those listed above) that, in the opinion of the investigator, precludes full participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Excess limb volume change | Baseline and 12 months after treatment
  Change in % of (excess) limb volume in the intervention group relative to control group

SECONDARY OUTCOMES:
LLIS survey | Baseline and 12 months after treatment
  Lymphedema-specific instrument to measure impairments, activity limitations, and participation restrictions in those living with any extremity lymphedema
L-Dex bioimpedance spectroscopy. | Baseline and 12 months after treatment
  Change in the Lymphedema Index (L-Dex) in the intervention group relative to control group. The L-Dex score has the requisite sensitivity and specificity to detect the differences in retained interstitial fluid that might discriminate the therapeutic responses of the treated patients. It has been established that the normal range of the L-Dex score is in the interval from -10 to +10 units; the higher score the more difference is in the retained interstitial fluid between the affected and unaffected limbs.
Histology | Baseline and 12 months after treatment
  Change in cutaneous histological architecture. The impact of treatment on the cutaneous histopathology will be evaluated through the use of an empirically derived scoring system and will be performed by a dermatopathologist.
ICG fluorescence imaging | Baseline and 12 months after treatment
  Change in lymphatic function assessed by ICG fluorescence imaging

CONTACTS AND LOCATIONS:
Overall Officials: David W Chang, MD, FACS, Principal Investigator — The University of Chicago Medicine & Biological Sciences; Rebecca Garza, MD, Study Director — The University of Chicago Medicine & Biological Sciences
Locations (2):
- United States (2):
  - The University of Chicago Biological Sciences Division/University of Chicago Medical Center, Chicago, Illinois
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang DW, Masia J, Garza R 3rd, Skoracki R, Neligan PC. Lymphedema: Surgical and Medical Therapy. Plast Reconstr Surg. 2016 Sep;138(3 Suppl):209S-218S. doi: 10.1097/PRS.0000000000002683. PMID 27556764
- [Background] Silva AK, Chang DW. Vascularized lymph node transfer and lymphovenous bypass: Novel treatment strategies for symptomatic lymphedema. J Surg Oncol. 2016 Jun;113(8):932-9. doi: 10.1002/jso.24171. Epub 2016 Feb 5. PMID 26846735
- [Background] Rochlin DH, Inchauste S, Zelones J, Nguyen DH. The role of adjunct nanofibrillar collagen scaffold implantation in the surgical management of secondary lymphedema: Review of the literature and summary of initial pilot studies. J Surg Oncol. 2020 Jan;121(1):121-128. doi: 10.1002/jso.25576. Epub 2019 Jun 18. PMID 31209884
- [Background] Inchauste S, Zelones J, Rochlin D, Nguyen DH. Successful treatment of lymphedema in a vasculopath and neuropathic patient. J Surg Oncol. 2020 Jan;121(1):182-186. doi: 10.1002/jso.25590. Epub 2019 Jun 22. PMID 31228351
- [Background] Garza RM, Ooi ASH, Falk J, Chang DW. The Relationship Between Clinical and Indocyanine Green Staging in Lymphedema. Lymphat Res Biol. 2019 Jun;17(3):329-333. doi: 10.1089/lrb.2018.0014. Epub 2018 Dec 18. PMID 30562150